CLINICAL TRIAL: NCT06167057
Title: Single Bladder Instillation With Chemotherapy Following Endoscopic Treatment for Upper Tract Urothelial Carcinoma to Reduce Bladder Recurrence
Brief Title: POST URS Chemotherapy Instillation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Yuval Freifeld, Head of Urologic-Oncology unit, Carmel Medical Center, Carmel Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0154-22-CMC-C
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: UTUC
Keywords: diagnostic URS; single-dose chemotherapy bladder instillation; IVR
MeSH Terms: interventions — Mitomycin; Gemcitabine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Multicenter, double arm, single blinded randomized trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental): Single post-operative MMC 40mg or gemcitabine 2gr in Saline 0.9% 50cc bladder instillation
  Interventions: Drug: Mitomycin/Gemcitabine
- B (Placebo Comparator): Single post-operative 50cc Saline 0.9% bladder instillation
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Mitomycin/Gemcitabine — UTUC treatment
  Arms: A
Drug: Saline — UTUC treatment
  Arms: B

SUMMARY:
The goal of this study is to evaluate the safety and oncological outcomes of single chemotherapy bladder instillation following endoscopic treatment for UTUC in UTUC suspected patients .The main aim is to determine the efficacy of a single, post URS, chemotherapy bladder instillation to reduce IVR.

Participants will be given single chemotherapy bladder instillation within 24h following ureteroscopy and will follow routine follow-up for IVR which will include white light cystoscopy ;patients with suspected IVR (based on either imaging or cystoscopy) will undergo TURBT.

DETAILED DESCRIPTION:
URS is routinely used for both diagnosis and treatment of UTUC - it is used either as an initial diagnostic procedure or as a curative procedure in cases amenable for endoscopic tumor ablation; either with low-risk disease or an imperative indication due to impaired renal function.

Following extirpative surgery patients are prone to IVR. Those patients undergo routine follow-up with cystoscopy and in cases of IVR require TURBT and further management based on bladder cancer protocols. In this setting, a single post-operative bladder instillation with various chemotherapeutic agents has shown a significant reduction in IVR rates following RNU.

Retrospective evidence suggests there is an increase IVR rates following URS for UTUC.

In this study the investigators seek to evaluate the efficacy of a single, post URS, bladder instillation with chemotherapy to reduce IVR.

ELIGIBILITY:
Inclusion Criteria:

* Radiographic and/or cytological suspicion for UTUC
* Planned endoscopic procedure for treatment / diagnosis of UTUC
* Patients with bladder cancer history are eligible if meeting both following criteria:

No recurrence within the last two years Are not on active bladder irrigation protocol

* Patients with history of UTUC are eligible if last endoscopic treatment or RNU was >1 year prior to enrollment
* Age ≥ 18 years
* Performance status ECOG 0-2

Exclusion Criteria:

* Subjects who have had bladder / prostate radiotherapy
* Subjects with bladder cancer history on active bladder irrigation protocols or with active disease within two years prior to enrollment
* Subjects with previously treated UTUC within one year prior to enrollment
* Subjects with metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2028-01-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
1 year IVR free survival | 1 year
  no intravesical recurrence of Upper Tract Urothelial Carcinoma in a patient for 1 year

SECONDARY OUTCOMES:
2 years IVR free survival | 2 years
  no intravesical recurrence of Upper Tract Urothelial Carcinoma in a patient for second year
Disease free survival | 2 years
High grade (>3) adverse events | 2 years
  Adverse events that are severe or medically significant but not immediately life threatening

CONTACTS AND LOCATIONS:
Locations (10):
- Israel (10):
  - Assuta Ashdod Hospital, Ashdod
  - Soroka University Medical Center, Beersheba
  - Shamir Medical Center, Be’er Ya‘aqov
  - Bnai Zion Medical Center, Haifa
  - Carmel Medical Center, Haifa
  - Rambam Health Care Campus, Haifa
  - Rabin Medical Center - Beilinson and Hasharon, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Ziv Medical Center, Safed
  - Tel Aviv Sourasky Medical Center - Ichilov, Tel Aviv

IPD SHARING:
Plan to Share IPD: No